CLINICAL TRIAL: NCT03707132
Title: Tourniquet on the Low Segment of the Uterus Reduces Blood Loss in Postpartum Hemorrhage During Hysterectomy for Placenta Accreta: Old But Gold
Brief Title: Tourniquet Reduces Blood Loss in Postpartum Hemorrhage During Hysterectomy for Placenta Accreta
Status: Completed | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, clinical associate professor, University Tunis El Manar
Other Study IDs: Garrot-Accreta
Record Dates: First submitted 2018-10-07; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Placenta Accreta; Post Partum Hemorrhage; Blood Loss Massive
Keywords: Tourniquet; low uterus segment; placenta accreta; hysterectomy; massive blood loss management
MeSH Terms: conditions — Placenta Accreta; Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tourniquet Group: 'Tourniquet: Folley catheter in the low segment of the uterus
  Interventions: Procedure: Tourniquet: Folley catheter in the low segment of the uterus
- Control Group: Standard hysterectomy is performed

INTERVENTIONS:
Procedure: Tourniquet: Folley catheter in the low segment of the uterus
  Groups: Tourniquet Group

SUMMARY:
Monocentric prospective observational study comparing the use of tourniquet in low uterus segement versus standard procedure in hysterectomy owing to placenta accreta

DETAILED DESCRIPTION:
It is a monocentric prospective observational case-control study in the Department "C" of Gynecology and Obstetrics in the Maternity and Neonatology Center of Tunis during three years from October 2014 to September 2017.

All parturient were informed about the possibility of performing a hysterectomy if accretization was clinically confirmed preoperatively. After obtaining written formal consent. all patients who underwent scheduled or emergency cesarean section for placenta accreta were included. Either it was highly suspected or confirmed by obstetrical imaging. MRI was always performed in cases of scheduled cesarean delivery. However, in cases of delayed transfer or if parturient was already in labor, only ultrasonography was done and considered as sufficient. Delivery was usually scheduled at 36 weeks of gestation.

Patients were allocated into two group: Group TG in which a tourniquet was systematically applied on the lower segment of the uterus during emergent hysterectomy, control group CG when the emergent caesarian hysterectomy was performed without a tourniquet. Allocation depended on the technique and the decision of the surgeon in charge.

After appropriate conditioning and monitoring, the cesarean section was performed under general anesthesia. The laparotomy was performed through a mid-line incision from the umbilicus to the pubic symphysis. Hysterotomy was made far from the placental insertion which was previously located by ultrasonography. The accretization was clinically checked immediately after delivery but no attempt was made to manually remove the placenta. The umbilical cord was ligated to its insertion and the uterus was quickly sutured with the placenta kept in place. Careful detachment of the bladder-uterus peritoneum was then carried out in order to lower the bladder and reduce the risk of bladder wounds. Tourniquet application procedure is described as following

1. Suturing hysterotomy with placenta kept in place.
2. After a cautious dissection a Folley catheter is placed in the lower segment of the uterus as tourniquet.
3. complete hysterectomy

ELIGIBILITY:
Inclusion Criteria:

* . All patients undergoing scheduled or emergency cesarean section for placenta accreta

Exclusion Criteria:

* No signs of accretetization upon artificial delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female pregnant subject
Study Population: All parturients with suspected placenta accreta either on MRI if the C section is scheduled or on Ultrasound if an emmergent delivery is set
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | peroperatively
  Blood spoliation during procedure
Hemoglobin variation | First 24 hours
  the differnece between the Baseline concentration of Hemoglobin and the lowest hemoglobin concentration noted during the procedure
Transfusion requirements | First 24 hours
  Number of red blood cells units transfused
procedure duration | peroperatively
  Time needed to perform hysterectomy from incision to skin closure
Intensive care transfer rate | first 24 hours
  Intensive care transfer following hysterectomy for placenta accreta

SECONDARY OUTCOMES:
length of stay in ICU | time from surgery up to 30 days postoperative
  duration of the stay in the ICU following hysterectomy for placenta accreta
clotting disorders | time from surgery up to 30 days postoperative
  Assessed by the incidence of Intravascular disseminated coagulopathy
Bladder wound | time from surgery up to 30 days postoperative
  Incidence of accidental bladder damage
Digestive wound | time from surgery up to 30 days postoperative
  Incidence of accidental digestive lesion

CONTACTS AND LOCATIONS:
Overall Officials: Hayen Maghrebi, Professor, Study Chair — Tunis Maternity Center

IPD SHARING:
Plan to Share IPD: Undecided